CLINICAL TRIAL: NCT07193160
Title: A Multicenter, Single-arm, Phase II Clinical Study of Sacituzumab Tirumotecan in Combination With Furmonertinib as Second-line Treatment for EGFR-mutant Advanced or Metastatic NSCLC After Failure of First-line Third-generation EGFR-TKI Therapy
Brief Title: Sacituzumab Tirumotecan in Combination With Furmonertinib as Second-line Treatment for EGFR-mutant Advanced or Metastatic NSCLC After Failure of First-line Third-generation EGFR-TKI Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-010
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: NSCLC; EGFR-mutant; ADC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sac-TMT + Furmonertinib (Experimental)
  Interventions: Drug: Sacituzumab Tirumotecan; Drug: Furmonertinib

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan — fixed dosage 4mg/kg iv, D1, D15, each 4 weeks one cycle. Drug reduction will be implemented according to the research plan.
  Other Names: sac-TMT; SKB264; MK-2870
Drug: Furmonertinib — 160mg QD or 80mg QD, each 4 weeks one cycle, according to the safety run-in phase, until confirmed by the investigator as imaging disease progression, intolerable toxicity, subject's request to terrminate treatment, or other treatment termination criteria specified in the protocol. Drug reduction will be implemented according to the research plan.

SUMMARY:
This study is a multicenter, single-arm, phase II clincial trial. The main objective of the study is to evaluate the efficacy and safety of the combination of Sacituzumab Tirumotecan (sac-TMT) and Furmonertinib in the treatment of EGFR-mutant advanced or metastatic NSCLC after failure of first-line Third-generation EGFR-TKI therapy.

DETAILED DESCRIPTION:
Monotherapy with third-generation EGFR-TKIs has become the standard first-line treatment for advanced NSCLC with EGFR mutations. However, acquired resistance inevitably occurs. ADCs harness the precise targeting and selectivity of monoclonal antibodies while capitalizing on the potent cytotoxic effects of their payload, thereby minimizing off-target toxicity. Sacituzumab Tirumotecan (sac-TMT) is a novel TROP2-directed ADC, had shown encouraging antitumor efficacy in previously treated patients with EGFR mutated advanced NSCLC. Theoretically, combination with small molecule inhibitors (including EGFR-TKI) are one of the combinational strategies for TROP2-ADC with synergistic mechanism.

This study aims to evaluate the efficacy and safety of furmonertinib plus Sacituzumab Tirumotecan in patients with EGFR mutated advanced NSCLC after failure of first-line third-generation EGFR-TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 to 75 years at the time of signing the informed consent form, regardless of gender; 2. Histologically or cytologically confirmed non-squamous NSCLC, which is locally advanced (Stage ⅢB/ⅢC) or metastatic (Stage Ⅳ) NSCLC that is not suitable for radical surgery and/or radical radiotherapy (whether concurrent chemotherapy is administered or not) [according to the 8th Edition of the Lung Cancer TNM Staging System by the Union for International Cancer Control (UICC) and the American Joint Committee on Cancer (AJCC)]; 3. There must be medical records showing evidence of previous EGFR mutation test results (known presence of EGFR mutations sensitive to EGFR-TKI [Ex19del, L858R], which may exist alone or concurrently with other EGFR mutations, possibly including T790M); 4. Subjects who experienced extracranial radiological progression after achieving remission (CR or PR) or stable disease (SD ≥ 6 months) during the first-line treatment with third-generation EGFR-TKI, but have not received further subsequent treatment (for subjects who received first-line treatment with a third-generation EGFR-TKI other than furmonertinib, the interval between the last dose of the first-line third-generation EGFR-TKI and the first dose of this study must be at least 8 days); 5. The brain metastasis status of subjects at enrollment must meet one of the following conditions:

  1. No brain metastasis;
  2. Stable brain metastasis, defined as no central nervous system (CNS) symptoms; or clinically stable for at least 4 weeks before enrollment, with all CNS symptoms returned to the baseline state; no evidence of new or enlarged brain metastatic lesions; and no need for treatment with glucocorticoids or anticonvulsants for at least 2 weeks before enrollment; 6. According to RECIST v1.1, the investigator assesses that there is at least one measurable target lesion that has not been irradiated, is non-central nervous system, and is measurable (if a subject has only one measurable lesion and must undergo tissue biopsy, the baseline tumor assessment needs to be performed at least 14 days after the screening biopsy); 7. Eastern Cooperative Oncology Group (ECOG) Performance Status Score (see Appendix 1 for details) of 0 or 1;

Exclusion Criteria:

* 1. Tumor histologically or cytologically confirmed to be combined with small cell lung cancer, neuroendocrine carcinoma, carcinosarcoma components, or squamous cell carcinoma components; 2. Radiologically diagnosed central nervous system (CNS) progression that occurred during or after previous first-line treatment with third-generation EGFR-TKI; 3. Subjects with known meningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or active central nervous system (CNS) metastasis; 4. Subjects who have previously received systemic antineoplastic therapy (such as chemotherapy and immunotherapy) for locally advanced or metastatic non-squamous NSCLC other than third-generation EGFR-TKI; 5. Previous treatment with TROP2-targeted therapy or any drug therapy targeting topoisomerase Ⅰ, including antibody-drug conjugate (ADC) therapy (including in the context of adjuvant or neoadjuvant therapy); 6. Radiotherapy with a total dose of > 30 Gy administered to lung lesions within 6 months before the first dose; non-thoracic radiotherapy or extensive radiotherapy with a total dose of > 30 Gy administered within 4 weeks before the first dose; palliative radiotherapy for symptom control is allowed, but it must be completed at least 2 weeks before the first dose; 7. History of other malignant tumors within 3 years before the first dose (except for tumors cured by local treatment, such as cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, carcinoma in situ of the cervix, etc.);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  Objective Response Rate (ORR) assessed according to the evaluation criteria for the efficacy of RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From treatment administration up to a maximum duration of 12 months.
  The time from the beginning of the patient's treatment to the disease progression or death for any reason. Based on RECIST v1.1.
Duration of Response (DoR) | Through study completion, an expected average of 12 months.
  The time from the first time the evaluation results meet CR or PR criteria to the observation of PD or death.
Disease Control Rate (DCR) | From treatment administration up to a maximum duration of 12 months.
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects after the last subject participating in.
Overall Survival (OS) | From treatment administration up to a maximum duration of 12 months.
  Time from start of treatment to death due to any cause.